CLINICAL TRIAL: NCT01622335
Title: Effect OF Nitrous Oxide On Acute Pain and Opioid Consumption, and Chronic
Brief Title: Effect OF Nitrous Oxide On Acute Pain and Opioid Consumption, and Chronic Pain After Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated per Principal Investigator decision.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Principal Investigatgor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1491-952
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Hysterectomy (& Wertheim); Nitrous Oxide; General Anesthesia
MeSH Terms: interventions — Nitrous Oxide; Anesthesia, General; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia with oxygen (Placebo Comparator): General anesthesia and Air
  Interventions: Other: General anesthesia with oxygen
- nitrous oxide and general anesthesia (Experimental): General anesthesia with Nitrous Oxide
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — General anesthesia with Nitrous Oxide, 70%, O2 30%) 1-5 L, Sevoflurane 1-2%, ETCO2: 32-35 mmHg.
  Arms: nitrous oxide and general anesthesia
Other: General anesthesia with oxygen — General anesthesia with(Air, 70%, O2 30%) 1-5 L, Sevoflurane 1-2%, ETCO2: 32-35 mmHg.
  Arms: General anesthesia with oxygen

SUMMARY:
The study is prospective and double blind. In the clinic, patients undergoing hysterectomy that meet the criteria for inclusion into the study and agreed to participate in the study will be randomized into two groups.

DETAILED DESCRIPTION:
The study is prospective and double blind. In the clinic, patients undergoing hysterectomy that meet the criteria for inclusion into the study and agreed to participate in the study will be randomized into two groups. In the first group of patients will receive Nitrous Oxide and In the second group of patients will receive oxygen during the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old at time of the first procedure
* Female
* American Society of Anesthesiologists physical status I or II
* Hysterectomy undergoing the general anesthesia

Exclusion Criteria:

* Neuropathic disease
* Chronic opioid users
* Contraindication for Nitrous Oxide receive
* Consent will not be obtained patient
* Psychiatric disorders
* Current or recent drug abuse (within past 6 months).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Nitrous oxide and chronic pain | 30 days post operative
  The of the effect of 50% N20/50% O2 on post hysterectomy in prevention of chronic pain.
Nitrous oxide and opioid consumption | 4 hours post operative
  The effect of 50% N20/50% O2 on post hysterectomy in decrease of opioid consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Gulhane Military Medical Academy Hospital, Etlik, Ankara, Turkey (Türkiye)